CLINICAL TRIAL: NCT04665466
Title: Combined AngiograpHy-derived Fractional Flow Reserve and Pullback Pressure Gradient Assessment to Better Discriminate Coronary ARTery Disease PAtients Benefiting From PercuTaneous Coronary InTERventioN
Brief Title: Implication of Coronary Artery Disease Burden and Pattern in Ischemia-causing Vessels With PCI
Acronym: CHART-PATTERN
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZS-20201206
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: QFR≤0.80 vessels with PCI strategy and low PPG index
  Interventions: Device: Quantitative Flow Ratio derived PPG
- Group B: QFR≤0.80 vessels with PCI strategy and high PPG index
  Interventions: Device: Quantitative Flow Ratio derived PPG
- Group C: QFR≤0.80 vessels with conservative strategy
  Interventions: Device: Quantitative Flow Ratio derived PPG

INTERVENTIONS:
Device: Quantitative Flow Ratio derived PPG — From coronary angiographic images, QFR will be calculated and virtual pullback curve will be abstracted and PPG index will be calculated as:
  PPG index={MaxPPG20mm/△QFRvessel+(1-length with functional disease/Total vessel length) }/2.

SUMMARY:
Ischemia-guided revascularization is the cornerstone of contemporary management of coronary artery disease (CAD). Coronary physiological assessment is advocated in the catheter laboratory to guide percutaneous coronary intervention (PCI), and it is widely accepted that an FFR ≤ 0.80 is a good indicator for vessels to benefit from revascularization. Nevertheless, a significant proportion of PCI patients continue to experience adverse events related to both stented segment and/or residual or diffuse disease. Our group recently demonstrated the feasibility of pullback pressure gradient (PPG) derived from virtual Quantitative Flow Ratio (QFR) pullback curve, which is an index of atherosclerosis functional pattern and can be used to epitomize the pathophysiological pattern of CAD as focal or diffuse.

In this regard, the current study will investigate the incremental value of PPG added to QFR haemodynamic assessment in ischemia-causing vessels received PCI in predicting adverse outcomes.

DETAILED DESCRIPTION:
Ischemia-guided revascularization is the cornerstone of contemporary management of coronary artery disease (CAD). Coronary physiological assessment is advocated in the catheter laboratory to guide percutaneous coronary intervention (PCI), and it is widely accepted that an FFR ≤ 0.80 is a good indicator for vessels to benefit from revascularization. Nevertheless, a significant proportion of PCI patients continue to experience adverse events related to both stented segment and/or residual or diffuse disease. Our group recently demonstrated the feasibility of pullback pressure gradient (PPG) derived from virtual Quantitative Flow Ratio (QFR) pullback curve, which is an index of atherosclerosis functional pattern and can be used to epitomize the pathophysiological pattern of CAD as focal or diffuse.

In this regard, the current study will investigate the incremental value of PPG added to QFR haemodynamic assessment in ischemia-causing vessels received PCI in predicting adverse outcomes.

The study cohort is derived from the PANDA-III study (Comparison of BuMA eG Based BioDegradable Polymer Stent With EXCEL Biodegradable Polymer Sirolimus-eluting Stent in "Real-World" Practice) (NCT02017275). In this cohort, vessels with measurable QFR≤ 0.80 will be included. According to the PPG index calculated from QFR virtual pullback curve and treatment strategy chosen, the included vessels were divided into three groups(vessels with PCI strategy and low PPG index (group A), vessels with PCI strategy with high PPG index (group B) and vessels with conservative strategy (group C)) and 2-year clinical outcomes for each group will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one vessel with measurable QFR≤ 0.80;
* PPG index can be calculated from virtual QFR pullback curve;
* The patient is willing to comply with specified follow-up evaluations;
* Patients who agree to accept the follow-up visits.

Exclusion Criteria:

* Culprit vessels for ACS myocardial infarction;
* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure;
* Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, stainless steel alloy, cobalt chromium, rapamycin, styrene-butylenes-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately pre-medicated;
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1003 patients with 1444 target vessels with measurable QFR≤ 0.80 from the PANDA-III study (Comparison of BuMA eG Based BioDegradable Polymer Stent With EXCEL Biodegradable Polymer Sirolimus-eluting Stent in "Real-World" Practice) (NCT02017275).
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Vessel-oriented composite outcome | at 2 years from index procedure
  Vessel-oriented composite outcome (VOCO) including vessel related ischemia-driven target vessel revascularization, vessel-related myocardial infarction (MI), and cardiac death.

SECONDARY OUTCOMES:
Cardiac death or vessel-related MI | at 2 years from index procedure
  Cardiac death or vessel-related MI
Vessel-related MI | at 2 years from index procedure
  Vessel-related MI
Cardiac death | at 2 years from index procedure
  Cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University; Bo Xu, MBBS, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu B, Gao R, Yang Y, Cao X, Qin L, Li Y, Li Z, Li X, Lin H, Guo Y, Ma Y, Wang J, Nie S, Xu L, Cao E, Guan C, Stone GW; PANDA III Investigators. Biodegradable Polymer-Based Sirolimus-Eluting Stents With Differing Elution and Absorption Kinetics: The PANDA III Trial. J Am Coll Cardiol. 2016 May 17;67(19):2249-2258. doi: 10.1016/j.jacc.2016.03.475. PMID 27173037